CLINICAL TRIAL: NCT07359287
Title: Impact of a Multimodal Intervention on Antibiotic Prescribing for Respiratory Infections in Primary Care: A Cluster-Randomized Trial
Brief Title: Impact of a Multimodal Intervention on Antibiotic Prescribing for Respiratory Infections in Primary Care
Acronym: GRASP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-0171
Record Dates: First submitted 2025-12-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-12

CONDITIONS: Angina; Acute Bronchiolitis; Acute Bronchitis; COPD Exacerbation (AECOPD); Laryngitis; Acute Otitis Media (AOM); Serous or Congestive Otitis; Viral Respiratory Infection (e.g., Influenza); Community-Acquired Pneumonia (CAP); Rhinitis / Nasopharyngitis; Acute Sinusitis
Keywords: Upper respiratory tract infection; Lower respiratory tract infection
MeSH Terms: conditions — Angina Pectoris; Bronchitis; Laryngitis; Otitis Media; Influenza, Human; Community-Acquired Pneumonia; Rhinitis; Nasopharyngitis; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The primary care practices in the control group do not receive any intervention and continue patient management according to their usual practices.
- Intervention group (Experimental): For the intervention group, two planned interventions will be planed and applied to the primary care practices:
  1. Use of the OPIV (Viral Infection Prescription Tool).
  2. A multidisciplinary collaboration protocol between general practitioners and pharmacists to evaluate antibiotic treatment durations. This intervention aims to strengthen collaborative practices. If a prescribed duration does not comply with recommendations, the pharmacist will discuss it with the prescriber, and the duration will be adjusted accordingly."
  Interventions: Other: Antibiotic prescribing according to guidelines

INTERVENTIONS:
Other: Antibiotic prescribing according to guidelines — If necessary, the general practitioner prescribes antibiotics to patients consulting for an upper or lower respiratory tract infection, according to the guidelines.
  Arms: Intervention group

SUMMARY:
Antimicrobial resistance (AMR), considered one of the greatest global threats by the WHO, justifies the development of initiatives to promote appropriate antibiotic use-especially in primary care, where most antibiotics in France are prescribed and where misuse remains common.

We are proposing a cluster-randomized controlled trial to evaluate the effectiveness of a bimodal intervention combining: (1) improved communication about the circulation of respiratory viruses, and (2) strengthened collaborative practices between general practitioners and pharmacists through a multidisciplinary protocol aimed at verifying that prescribed treatment durations comply with guidelines.

The study will include six primary care practices (24 physicians), with three practices in each study arm.

The aim of this project is to assess whether the bimodal intervention can reduce the duration of antibiotic treatments for upper and lower respiratory tract infections. The first component (a "viral infection prescription" tool) focuses on reducing unnecessary treatment initiation, while the second (pharmacist-led review) aims to shorten excessive prescription durations.

ELIGIBILITY:
Inclusion Criteria:

- Patient seen in consultation for an upper or lower respiratory tract infection (Angina, Acute bronchiolitis, Acute bronchitis, COPD exacerbation (AECOPD), Laryngitis, Acute otitis media (AOM), Serous or congestive otitis, Viral respiratory infection (e.g., influenza), Community-acquired pneumonia (CAP), Rhinitis / Nasopharyngitis, Acute sinusitis)

Exclusion Criteria:

- Patient under legal protection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4500 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of antibiotic treatment days prescribed for upper and lower respiratory tract infections. | The primary outcome is measured at the time of prescription (i.e. at the baseline)
  The primary outcome of the study will be the number of antibiotic treatment days prescribed for upper and lower respiratory tract infections. This outcome is a composite measure reflecting the impact of both interventions. Antibiotic duration will be assessed by running a query in the electronic medical record system of the participating primary care practices. The primary outcome will be evaluated at the baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU CAEN Normandie, Caen, France

IPD SHARING:
Plan to Share IPD: No